CLINICAL TRIAL: NCT05174286
Title: Community Health Workers United to Reduce Colorectal Cancer and Cardiovascular Disease Among People at Higher Risk
Acronym: CHURCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Olajide Williams, Professor of Neurology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT9307; 1P50MD017341 (NIH)
Record Dates: First submitted 2021-11-05; First posted 2021-12-30 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: Community Health Workers; Colorectal Cancer; Cardiovascular Disease; Screening; Prevention
MeSH Terms: conditions — Colorectal Neoplasms; Cardiovascular Diseases | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Screening, Brief Intervention, and Referral to Treatment (SBIRT) (Experimental): Participants randomized to this arm will receive:
  1. SBIRT is an evidence-based approach originally designed for people at risk of developing mental disorders. SBIRT is composed of three components: Screening with a validated instrument, Brief Intervention, Referral to Treatment. Motivational Interviewing (MI) is an empirically tested, person-centered, behavior change intervention designed to guide, elicit, and strengthen motivation for change. It decreases ambivalence and increases motivation for treatment.
  2. Culturally-adapted Alive! Program, which is a cost-effective, lifestyle coaching web-based automated platform that includes step-by-step individualized tailoring, feedback, and weekly guidance through interactive emails focused on increasing physical activity, improving eating habits, and weight control.
  Interventions: Behavioral: SBIRT
- Referral as Usual (RAU) (Active Comparator): Participants randomized to this arm will receive Referral as Usual (RAU), which will involve distributing CRC health educational materials (e.g. NCI or Centers For Disease Control brochures that include new guidelines) and contact information for screening service providers in our target community.
  Interventions: Behavioral: Referral as Usual (RAU)

INTERVENTIONS:
Behavioral: SBIRT — SBIRT is an evidence-based approach originally designed for people at risk of developing mental disorders. SBIRT is composed of three components: Screening with a validated instrument, Brief Intervention, Referral to Treatment. Motivational Interviewing (MI) is an empirically tested, person-centered, behavior change intervention designed to guide, elicit, and strengthen motivation for change. It decreases ambivalence and increases motivation for treatment.
  The investigators will utilize the Culturally-adapted Alive! Program - a cost-effective, lifestyle coaching web-based automated platform that includes step-by-step individualized tailoring, feedback, and weekly guidance through interactive emails focused on increasing physical activity, improving eating habits, and weight control.
  Other Names: Culturally-adapted ALIVE! Program (CAP)
  Arms: Screening, Brief Intervention, and Referral to Treatment (SBIRT)
Behavioral: Referral as Usual (RAU) — Referral as Usual will involve distributing CRC health educational materials (e.g. NCI or CDC brochures that include new guidelines) and contact information for screening service providers in our target community.
  Arms: Referral as Usual (RAU)

SUMMARY:
The overall goal of this study is to develop a comprehensive, culturally tailored community-based colorectal cancer (CRC) prevention model with a dual emphasis on reducing CRC risk along with its CVD risk factors. The study intervention has two components: Screening, Brief Intervention, and Referral to Treatment (SBIRT) to address CRC screening and a web-based lifestyle program called "Alive!" to address CVD risk factors linked to CRC. The C.H.U.R.C.H. Trial (Community Health workers (CHW) United to Reduce Colorectal cancer and cardiovascular disease among people at Higher risk) has four specific aims: (1) to compare the effect of a CHW-Led SBIRT (Intervention) to Referral As Usual (RAU) (Usual Care) on guideline-concordant CRC screening uptake; (2) to evaluate the effect of a Culturally Adapted CHW-linked Alive! (CACA) program incorporated into the intervention arm on dietary inflammatory score (DIS); (3) to evaluate the effect of CACA on changes in Life Simple-7 (LS7) scores; and (4) to examine the multi-level contextual mechanisms and factors influencing CHW effectiveness, reach, and implementation of CRC screening uptake and CACA activities through a mixed-methods process evaluation. Given the broad reach and influence of churches, results from this study can be used to inform future scale up of this multi-pronged intervention.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most lethal cancer in the U.S with the highest incidence and mortality rates among African Americans (AAs) compared to other racial groups. Despite these disparities, which includes premature mortality, AAs are the least likely to undergo CRC screening, have precancerous colorectal polys removed, and have CRC detected at stages early enough for curative excision. Lower screening rates are linked to the downstream effects of structural inequities such as access to care, knowledge of screening options and benefits, health system mistrust, fear and anxiety. Although reducing the burden of CRC is best accomplished by screening, compelling evidence links inflammatory diets and cardiovascular disease (CVD) risk factors to increased CRC risk. This proposal aims to develop a community-based prevention model to reduce CRC and cardiovascular disease (CVD) risk among AAs.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking
2. Aged 45 years and older
3. Not up-to-date with CRC
4. Working telephone
5. Can provide informed consent

Exclusion Criteria:

1. Non-English speaking
2. <45 years old

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2023-03-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
CRC Screening Uptake | 6 months post-screening
  Screening uptake (clinic-based colonoscopy or home-based stool test) (Primary Outcome) is the subject's self-report of completing a CRC screening test plus the research team's verification of this completion from medical records.

SECONDARY OUTCOMES:
Change in Dietary Inflammatory Score (Dietary Screening Measure) | Baseline and 6 months post-screening
  Assessment of participant eating habits via the culturally-adapted ALIVE! program will be captured by the Block Food Frequency Questionnaire (FFQ) that generates the dietary inflammatory score (DIS) which can be used to examine associations between inflammatory diets, cardiovascular diseases and colorectal cancer.
Change in Life's Simple 7 Score (CVD Risk Screening Measure) | Baseline, 6 months post-screening and 1 year post-screening
  Evaluation of CVD risk factors using the Life Simple-7 (LS7) measure. LS7 scores range from 0 to 14 and are calculated from the composite of the factor scores. CVD health is then classified as inadequate (0-4), average (5-9), or optimum (10-14). Achieving a greater number of ideal LS7 metrics is associated with lower risk of dying after stroke and all cause cardiovascular mortality in a dose dependent manner.

CONTACTS AND LOCATIONS:
Overall Officials: Olajide A. Williams, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through submission of study findings to peer-reviewed journals. De-identified data will also be shared at community forums and academic conferences.
Supporting Information: Study Protocol
Time Frame: Data will be available six months after publication in a peer-reviewed journal article.
Access Criteria: The study Investigators, Dr. Olajide Williams, will create criteria and review requests for data sharing access. Data will be available to analyze types of clinical and demographic factors impact study outcomes.

REFERENCES:
- [Background] Jackson CS, Oman M, Patel AM, Vega KJ. Health disparities in colorectal cancer among racial and ethnic minorities in the United States. J Gastrointest Oncol. 2016 Apr;7(Suppl 1):S32-43. doi: 10.3978/j.issn.2078-6891.2015.039. PMID 27034811
- [Background] De Jesus M, Puleo E, Shelton RC, McNeill LH, Emmons KM. Factors associated with colorectal cancer screening among a low-income, multiethnic, highly insured population: does provider's understanding of the patient's social context matter? J Urban Health. 2010 Mar;87(2):236-243. doi: 10.1007/s11524-009-9420-1. Epub 2009 Dec 31. PMID 20043214
- [Background] Sly JR, Edwards T, Shelton RC, Jandorf L. Identifying barriers to colonoscopy screening for nonadherent African American participants in a patient navigation intervention. Health Educ Behav. 2013 Aug;40(4):449-57. doi: 10.1177/1090198112459514. Epub 2012 Oct 19. PMID 23086556
- [Background] Lumpkins CY, Coffey CR, Daley CM, Greiner KA. Employing the church as a marketer of cancer prevention: a look at a health promotion project aimed to reduce colorectal cancer among African Americans in the Midwest. Fam Community Health. 2013 Jul-Sep;36(3):215-23. doi: 10.1097/FCH.0b013e31829159ed. PMID 23718957
- [Background] Maxwell AE, Lucas-Wright A, Santifer RE, Vargas C, Gatson J, Chang LC. Promoting Cancer Screening in Partnership With Health Ministries in 9 African American Churches in South Los Angeles: An Implementation Pilot Study. Prev Chronic Dis. 2019 Sep 19;16:E128. doi: 10.5888/pcd16.190135. PMID 31538568
- [Background] Shelton RC, Thompson HS, Jandorf L, Varela A, Oliveri B, Villagra C, Valdimarsdottir HB, Redd WH. Training experiences of lay and professional patient navigators for colorectal cancer screening. J Cancer Educ. 2011 Jun;26(2):277-84. doi: 10.1007/s13187-010-0185-8. PMID 21287311
- [Derived] Williams O, Ting T, Matthews L, Block G, Block T, Teresi J, Eimicke J, Kong J, Silver S, Ravenell J, Mallaiah J, Jammalamadaka S, Nelson LM, Karmally W, Hankerson S. Community Health workers United to Reduce Colorectal cancer and cardiovascular disease among people at Higher risk (CHURCH): study protocol for a randomized controlled trial. Trials. 2024 Apr 26;25(1):283. doi: 10.1186/s13063-024-08110-z. PMID 38671470
- [Derived] Williams O, Ting T, Matthews L, Block G, Block T, Teresi J, Eimicke J, Kong J, Silver S, Ravenell J, Mallaiah J, Jammalamadaka S, Nelson LM, Karmally W, Hankerson S. Community Health workers United to Reduce Colorectal cancer and cardiovascular disease among people at Higher risk (CHURCH): study protocol for a randomized controlled trial. Res Sq [Preprint]. 2024 Apr 9:rs.3.rs-3797889. doi: 10.21203/rs.3.rs-3797889/v1. PMID 38659874